CLINICAL TRIAL: NCT02556697
Title: In Vivo Endomicroscopic Description of Pulmonary Microcirculation in Systemic Sclerosis and Emphysema Patients
Acronym: MiPECSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/093/HP
Record Dates: First submitted 2015-09-17; First posted 2015-09-22 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Disease; Pulmonary Emphysema
MeSH Terms: conditions — Lung Diseases; Pulmonary Emphysema | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with a suspicion of emphysema (Experimental): A bronchoscopy with in vivo confocal endomicroscopy is assessed for patient with a suspicion of emphysema
  Interventions: Device: Bronchoscopy with in vivo confocal endomicroscopy
- patients with a suspicion of scleroderma (Experimental): A bronchoscopy with in vivo confocal endomicroscopy is assessed for patient with a suspicion of sclerodermia
  Interventions: Device: Bronchoscopy with in vivo confocal endomicroscopy

INTERVENTIONS:
Device: Bronchoscopy with in vivo confocal endomicroscopy — A bronchoscopy with in vivo confocal endomicroscopy is done for patients with a suspicion of emphysema or for patients with a suspicion of scleroderma

SUMMARY:
Systemic sclerosis (SSc) is a generalized disorder of connective tissue, arterioles and microvessels, characterized by the occurrence of fibrosis and vascular obliteration phenomena. The alterations in lung microvessels are found in pulmonary involvement of scleroderma, which are the most serious complications of the disease.

In pulmonary emphysema, there are also changes in pulmonary microvasculature, which are involved in the onset and development of the disease.

The confocal endomicroscopy is an endoscopic technique which can be performed during a bronchoscopy. This technique makes it possible to observe in real time the most distal pulmonary elements at the microscopic scale. After injection of fluorescein, then the technique of observing the pulmonary microvasculature, in vivo and in situ.

The characterization of microvascular lesions in these two pathologies could improve understanding of their mechanisms and ultimately improve the early management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scleroderma with diffuse interstitial pneumonia, indicating a bronchoscopy.
* Patients with pulmonary emphysema indication for bronchoscopy.
* Age greater than 18 years.
* Having an affiliation to social security.
* Signed informed consent.

Exclusion Criteria:

* Severe chronic respiratory insufficiency against-indicating the completion of a bronchoscopy
* Hypercapnia defined by a PaCO2 ≥ 6 kPa
* Disorders of hemostasis against-indicating performing a bronchoscopy
* Anticoagulant therapy can not be interrupted time of completion of the examination
* A history of pneumonectomy or contralateral exploration in a nonfunctional lung
* Contraindication to the injection of fluorescein (including treatment with beta-blocker eye drops or po) or one of its excipients
* History of an injection poorly tolerated fluorescein
* A history of food allergy or drug known
* Myocardial infarction <1 month
* Unstable angina
* Pregnant or lactating woman, premenopausal women without adequate contraception
* Person under guardianship
* Patient participating in another trial / participating in another trial within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Measurement of extra-alveolar diameter of capillaries of patient with pulmonary emphysema or pulmonary scleroderma | Day 1
  Extra-alveolar diameter of capillaries is assessed using in vivo confocal endomicroscopy
Measurement of intercapillary distance of patient with pulmonary emphysema or pulmonary scleroderma | Day 1
  Intercapillary distance is assessed using in vivo confocal endomicroscopy
Measurement of length of the capillary portions of patient with pulmonary emphysema or pulmonary scleroderma | Day 1
  Length of the capillary is assessed using in vivo confocal endomicroscopy

SECONDARY OUTCOMES:
Measurement of alveolar diameter entries of patient with pulmonary emphysema or pulmonary scleroderma | Day 1
  Alveolar diameter entries is assessed using in vivo confocal endomicroscopy
Measurement of axial thickness of elastic fibers of patient with pulmonary emphysema or pulmonary scleroderma | Day 1
  Axial thickness of elastic fibers is assessed using in vivo confocal endomicroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu SALAUN, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France